CLINICAL TRIAL: NCT03892889
Title: A Phase IIIb Multi-Center, Open-Label, Mirror-Image, Trial in Adult Subjects With Schizophrenia Treated Prospectively for 6-months With Abilify MyCite®
Brief Title: A Trial in Adult Participants With Schizophrenia Treated Prospectively for 6-months With Abilify MyCite®
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: Study has stopped for having met the primary endpoint.
Sponsor: Otsuka Pharmaceutical Development & Commercialization, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Health Services Research
Other Study IDs: 031-201-00301
Record Dates: First submitted 2019-03-21; First posted 2019-03-27 (Actual); Results first posted 2021-09-05 (Actual); Last update posted 2021-09-05 (Actual); Status verified 2021-08

CONDITIONS: Schizophrenia
MeSH Terms: conditions — Schizophrenia

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: Yes | US Export: No

ARMS (1):
- Abilify MyCite® (Experimental): Participants received Abilify MyCite® a combination product of aripiprazole tablet embedded with sensor and wearable patch for 3 months (Months 1 to 3) and continued for an additional 3 months (Months 4 to 6) as per investigators assessment or switch to a standard-of-care treatment of oral atypical antipsychotics or a long acting injectable.
  Interventions: Combination Product: Abilify MyCite®

INTERVENTIONS:
Combination Product: Abilify MyCite® — Combination product of aripiprazole tablet embedded with sensor and wearable patch.

SUMMARY:
To compare inpatient psychiatric hospitalization rates while participants are on oral standard-of-care antipsychotic treatment and later switched to Abilify MyCite®.

DETAILED DESCRIPTION:
This study is designed to assess the difference between inpatient psychiatric hospitalization rates in participants on oral standard-of-care antipsychotic treatment(s) for a period of 6 months followed by a switch to Abilify MyCite® for a period of 3 months (Months 1 to 3).

At the Month 3 visit, the investigator should decide if participants will continue on Abilify MyCite® for an additional 3 months (Months 4 to 6) or switch to a standard-of-care treatment for the duration of treatment.

Participants must have had at least 1 inpatient psychiatric hospitalization within 4 years (48 months) and must have been prescribed oral antipsychotics for at least 6 months or longer prior to screening.

Participants will enter a screening period (up to 45 days). If deemed eligible to participate, participants will enter an open-label Abilify MyCite® treatment prospective phase for up to 6 months.

All participants who complete or withdraw from the trial while on Abilify MyCite® will receive a telephone call for safety follow-up approximately 30 days after their last trial visit.

The trial will be conducted at 75 sites in the United States, 493 participants will be screened in order to enroll 320 participants and complete 224 participants. There was an interim analysis planned for the study.

ELIGIBILITY:
Inclusion Criteria:

* Participants must be willing and able to give written informed consent, adhere to trial procedures and able to read and understand English.
* Male and female participants 18 to 65 years of age.
* Participants must possess a smartphone and is familiar with its use and is willing to download and interact with the Abilify MyCite® app. Participants with a smartphone, that is not compatible with the Abilify MyCite® app will be offered a loaner phone for the trial period.
* Clinical diagnosis of schizophrenia and able to ingest oral medication.
* Positive and Negative Syndrome Scale (PANSS) total score between 60-90.
* Participants currently prescribed oral atypical antipsychotic medication including aripiprazole or appropriate for aripiprazole treatment for 6 months or longer.
* Participants are required to have had an inpatient hospitalization for schizophrenia within the last 48 months prior to entering the trial.
* Skin on the anterior chest just above the lower edge of the rib cage that is free of any dermatological problems.

Exclusion Criteria:

* Females who are breast-feeding and/or who are pregnant.
* Sexually active males or women of childbearing potential (WOCBP) who do not agree to practice 2 different methods of birth control or remain abstinent during the trial and for 30 days after the last dose of Abilify MyCite®.
* Any participants who participated in another clinical trial within 30 days of enrollment.
* Participants who are currently being treated with an LAI antipsychotic or have been treated with an LAI in the retrospective 6-month phase.
* Participants with a current DSM-5 diagnosis other than schizophrenia.
* Participants with a known allergy to adhesive tape or any pertinent components of the patch or aripiprazole tablet embedded with an IEM sensor.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 277 (Actual)
Dates: Start 2019-04-29 (Actual); Primary Completion 2020-08-12 (Actual); Study Completion 2020-09-29 (Actual)

CONTACTS AND LOCATIONS:
Locations (68):
- United States (68):
  - Alea Research, Phoenix, Arizona
  - Woodland International Research Group, Little Rock, Arkansas
  - ADVANCED RESEARCH CENTER, Inc., Anaheim, California
  - CITrials, Bellflower, California
  - Synexus, Cerritos, California
  - CMB Clinical Trials, Colton, California
  - ProScience Research Group, Culver City, California
  - Collaborative Neuroscience Network, LLC, Garden Grove, California
  - Behavioral Research Specialists, LLC, Glendale, California
  - San Fernando Mental Health Center, Granada Hills, California
  - Om Research LLC, Lancaster, California
  - Synergy San Diego, Lemon Grove, California
  - CalNeuro Research Group, Los Angeles, California
  - Pacific Research Partners, Oakland, California
  - Excell Research, Inc, Oceanside, California
  - CNRI-Los Angeles, Pico Rivera, California
  - Prospective Research Innovations Inc., Rancho Cucamonga, California
  - CITrials, Riverside, California
  - CNRI-San Diego, LLC, San Diego, California
  - Artemis Institute for Clinical Research, San Diego, California
  - CITrials, Inc., Santa Ana, California
  - Siyan Clinical Research, Santa Rosa, California
  - Collaborative Neuroscience Network, LLC, Torrance, California
  - Sarkis Clinical Trials, Gainesville, Florida
  - Indago Research & Health Center, Inc., Hialeah, Florida
  - New Life medical Research Inc., Hialeah, Florida
  - Galiz Research, Hialeah, Florida
  - Innovative Clinical Research, Inc., Lauderhill, Florida
  - Premier Clinical Research Institute Inc., Miami, Florida
  - CCM Clinical Research Group, Miami, Florida
  - Prestige Clinical Research Center Inc., Miami, Florida
  - Stedman Clinical Tirlas, Tampa, Florida
  - Nova Psychiatry, Inc, Winter Park, Florida
  - Emory, Atlanta, Georgia
  - Synexus Clinical Research US, Atlanta, Georgia
  - iResearch Atlanta, Decatur, Georgia
  - iResearch Savannah, Savannah, Georgia
  - Uptown Research Institute, Chicago, Illinois
  - AMITA Health, Hoffman Estates, Illinois
  - SIU School of Medicine, Springfield, Illinois
  - Lake Charles Clinical Trial, Lake Charles, Louisiana
  - Michigan Clinical Research Institute, Ann Arbor, Michigan
  - Precise Research Centers, Flowood, Mississippi
  - Arch Clinical Trials, LLC, St Louis, Missouri
  - PsychCare Consultants Research, St Louis, Missouri
  - Alivation Research, LLC., Lincoln, Nebraska
  - Altea Research Institute, Las Vegas, Nevada
  - Kolade Research Institute/Cal Psychiatric Services, Las Vegas, Nevada
  - Hassman Research Institute, Berlin, New Jersey
  - Synexus US, Jamaica, New York
  - Manhattan Psychiatric Center, New York, New York
  - Manhattan Behavioral Medicine PLLC, New York, New York
  - Finger Lakes Clinical Research, Rochester, New York
  - Richmond Behavioral Associates, Staten Island, New York
  - Midwest Clinical Research Center, Dayton, Ohio
  - Signature Research Associates Inc, Fairlawn, Ohio
  - Charak Clinical research Center, Garfield Heights, Ohio
  - Neuro-Behavioral Clinical Research, Inc., North Canton, Ohio
  - The Rivus Wellness & Research Institute, Oklahoma City, Oklahoma
  - Cutting Edge Research Group, Oklahoma City, Oklahoma
  - Suburban Research Associates, Media, Pennsylvania
  - Psychiatric Consultants, PC, Franklin, Tennessee
  - Community Clinical Research, Inc., Austin, Texas
  - InSite Clinical Research, DeSoto, Texas
  - Baylor College of Medicine, Houston, Texas
  - Pillar Clinical Research, Richardson, Texas
  - Noetic Psychiatry, Springville, Utah
  - Northwest Clinical Research Center, Bellevue, Washington

IPD SHARING:
Plan to Share IPD: Yes
Anonymized Individual participant data (IPD) that underlie the results of this study will be shared with researchers to achieve aims pre-specified in a methodologically sound research proposal. Small studies with less than 25 participants are excluded from data sharing.
Supporting Information: Study Protocol, SAP, CSR
Time Frame: Data will be available after marketing approval in global markets, or beginning 1-3 years following article publication. There is no end date to the availability of the data.
Access Criteria: Otsuka will share data on an Otsuka-owned remotely accessible data sharing platform with Python and R analytical software. Research requests should be directed to clinicaltransparency@Otsuka-us.com
URL: https://clinical-trials.otsuka.com

REFERENCES:
- [Derived] Jan M, Coppin-Renz A, West R, Gallo CL, Cochran JM, Heumen EV, Fahmy M, Reuteman-Fowler JC. Safety Evaluation in Iterative Development of Wearable Patches for Aripiprazole Tablets With Sensor: Pooled Analysis of Clinical Trials. JMIR Form Res. 2023 Dec 12;7:e44768. doi: 10.2196/44768. PMID 38085556
- [Derived] Cohen EA, Skubiak T, Hadzi Boskovic D, Norman K, Knights J, Fang H, Coppin-Renz A, Peters-Strickland T, Lindenmayer JP, Reuteman-Fowler JC. Phase 3b Multicenter, Prospective, Open-label Trial to Evaluate the Effects of a Digital Medicine System on Inpatient Psychiatric Hospitalization Rates for Adults With Schizophrenia. J Clin Psychiatry. 2022 Apr 11;83(3):21m14132. doi: 10.4088/JCP.21m14132. PMID 35421287

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants took part in the study at 58 investigative sites in the United States from 29 April 2019 to 12 August 2020.
Pre-assignment Details: Participants who were on oral standard-of-care antipsychotic treatments for a period of 6 months prior to Baseline (Day 1) were assessed retrospectively and were enrolled in the Prospective Period on Day 1 to receive Abilify MyCite® for a period of 3 months (Months 1 to 3) and to continue with same treatment or standard of care up to Month 6.
Period: Overall Study
Arm/Group | Abilify MyCite®
Started | 277
Completed | 73
Not Completed | 204
Not completed — Adverse Event | 17
Not completed — Lack of Efficacy | 1
Not completed — Lost to Follow-up | 46
Not completed — Non-compliance with study drug | 22
Not completed — Pregnancy | 1
Not completed — Protocol Deviation | 3
Not completed — Withdrawal by Subject | 50
Not completed — Withdrawal by Caregiver | 1
Not completed — Study Terminated by Sponsor | 50
Not completed — Physician Decision | 8
Not completed — Reason not Specified | 5

BASELINE CHARACTERISTICS:
Population: Intent-to-Treat (ITT) Sample included all enrolled sample who met the study inclusion/exclusion criteria and who are intended to receive study medication in the Prospective Phase.
Arm/Group | Abilify MyCite®
Number analyzed (Participants) | 277
Age, Continuous [Mean (Standard Deviation); unit: Years] | 44.2 (12.4)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 95
  Male | 182
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 52
  Not Hispanic or Latino | 223
  Unknown or Not Reported | 2
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 4
  Asian | 5
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 167
  White | 98
  More than one race | 0
  Unknown or Not Reported | 3

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants With Inpatient Psychiatric Hospitalization
Description: Percentage of participants with inpatient psychiatric hospitalization in Prospective Period With at least one hospitalization in Retrospective Period.
Time Frame: Retrospective Period [Month -6 to Baseline (Day 1)] up to Prospective Period (Day 1 to Month 3)
Population: Modified Intent-to-Treat (mITT) Sample included data from all participants entering the prospective phase who have completed the first 3-months of dosing on Abilify MyCite®.
Measure: Number; unit: percentage of participants
Arm/Group | Abilify MyCite®
Number analyzed (Participants) | 113
percentage of participants | 0.0

2. Secondary Outcome: Percentage of Days With Improved Adherence
Description: Improved adherence was based on the overall proportion of days covered (PDC) in participants compliant with study drug administration in the Prospective period on Prospective Abilify MyCite® versus Retrospective Period on oral atypical antipsychotics. PDC was calculated as = number of days 'covered' in the Respective Period/number of days in the period * 100.
Time Frame: Retrospective Period [-1 to -3 months prior to Baseline (Day 1)] up to Prospective Period (1 to 3 months)
Population: ITT Sample included all enrolled sample who met the study inclusion/exclusion criteria and who are intended to receive study medication in the Prospective Phase. Overall number analyzed is the number of participants with confirmed retrospective prescription data to conduct the PDC calculation.
Measure: Mean (Standard Deviation); unit: percentage of days
Arm/Group | Abilify MyCite®
Number analyzed (Participants) | 162
percentage of days
  PDC in Retrospective Period | 51.0 (37.9)
  PDC in Prospective Period | 77.5 (31.8)
Statistical Analysis 1: Comparison: Abilify MyCite®; Test type: Other; p < 0.0001, paired t-test — Paired t-test was used based on the prospective phase efficacy sample when applicable

ADVERSE EVENTS:
Time Frame: Up to 6 months
Arm/Group | Abilify MyCite®
All-Cause Mortality (participants affected / at risk) | 1/277
Serious Adverse Events (participants affected / at risk) | 6/277
Other Adverse Events (participants affected / at risk) | 0/277
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Abilify MyCite® (N=277)
Pancreatitis Acute (Gastrointestinal disorders) | 1
Drug Hypersensitivity (Immune system disorders) | 1
Pneumonia Bacterial (Infections and infestations) | 1
Cerebrovascular Accident (Nervous system disorders) | 1
Schizophrenia (Psychiatric disorders) | 2

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Sponsor reserves the right to review results publications prior to public release and can delay such publications for a period greater than 60 days but no more than 120 days from the date that the publication is submitted to the Sponsor for review. Sponsor can require changes to the publication to protect Sponsor's intellectual property rights and/or confidential information and reserves the right to limit publication timing and scope of data published based on the number of study locations.

DOCUMENTS (2):
  • Study Protocol (2019-02-11): https://cdn.clinicaltrials.gov/large-docs/89/NCT03892889/Prot_000.pdf
  • Statistical Analysis Plan (2020-10-28): https://cdn.clinicaltrials.gov/large-docs/89/NCT03892889/SAP_001.pdf